CLINICAL TRIAL: NCT03559634
Title: Feasibility Trial of Hormonal Contraceptive Initiation Program in the Pediatric Emergency Department
Brief Title: Contraception Initiation Feasibility in the Pediatric ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201805104
Record Dates: First submitted 2018-05-22; First posted 2018-06-18 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Contraception; Contraception Behavior
MeSH Terms: conditions — Contraception Behavior | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Using an electronic application, participants answer survey questions about their sexual history, medical history, and contraceptive preferences. They will watch a video that overviews the types of hormonal contraception. Then, based on survey answers, they will be able to watch more in-depth educational videos on methods that they qualify for. Participants will only be offered methods that are considered low risk and without any contraindication based upon responses to survey screening. This may include, contraceptive implant, medroxyprogesterone acetate injection, microgestin pills, xulane patch, or intravaginal ring. Participants will then be given the opportunity to initiate contraception in the ED. All participants will be referred for follow up outpatient health services. Subjects who have medical contraindications to certain contraceptive medications will be given a standardized handout that explains why they were not eligible for the medication(s) while in the ED.
  Interventions: Diagnostic Test: Intervention Group
- Control Group (Other): Using an electronic application, participants answer survey questions about their background, sexual history, medical history, and contraceptive preferences. They will watch a video that overviews the types of hormonal contraception with brief pros and cons of each method. Then, based on participants medical history and contraceptive preferences they will be able to watch more in-depth counseling and educational videos on contraceptive methods that they qualify for. After these videos they will be given information on where they will be able to follow up to receive these contraceptive methods if they wish to start a method. Subjects who have medical contraindications to certain hormonal contraceptive medications will be given a standardized handout that explains why they were not eligible for the medication(s), should this come up in future discussions with their providers.
  Interventions: Other: Control Group

INTERVENTIONS:
Diagnostic Test: Intervention Group — The electronic application will collect screening health information and contraceptive preferences about the participant. Then, using branch logic, decide which contraceptive options the participant would qualify for based on health history answers. Contraceptive choices being offered include the contraceptive implant, injection, pill, patch, or ring. They will then be able to watch videos about methods they are eligible for. The participant can then decide if they would like to start a medication they qualify for in the ED.
  Arms: Intervention group
Other: Control Group — The electronic application will collect screening health information and contraceptive preferences about the participant. Then, using branch logic, decide which contraceptive options the participant would qualify for based on health history answers. This includes the contraceptive implant, injection, pill, patch, or ring. They will then be able to watch videos about methods they are eligible for. Participants will then be given follow up information on outpatient locations where they can receive these contraceptive methods.
  Arms: Control Group

SUMMARY:
Many female adolescents using the pediatric emergency department (ED) are at higher risk for unintended pregnancy. This is a significant public health issue and hormonal contraception is the mainstay of prevention. Many barriers to hormonal contraception exist and other studies have demonstrated that referral from the ED for hormonal contraception leads to poor follow up.

This study will be a pilot study to assess the feasibility of initiating hormonal contraception in the pediatric ED.

DETAILED DESCRIPTION:
This study will assess the feasibility of initiating hormonal contraception in the pediatric ED. Currently, all 15-21-year-old patients receiving care in our ED are asked to complete an adolescent heath questionnaire to identify risk-factors for sexually transmitted infections (STIs). Sexually active female patients who indicate on this questionnaire they are not currently using hormonal contraception will be eligible for participation in this study.

Potential participants will be screened using the EMR and eligible patients will be approached. Consent will be obtained from adults directly and from a parent or guardian for minors that have one present. For minors that present without a parent or guardian, assent only with be obtained from the minor. Participants will be randomized into two groups, an intervention group and a control group. Participants in both groups will be given tablet computer and, through a software application on the tablet, answer questions electronically about their background, medical history, and contraceptive preferences. They will then be shown a video that provides an overview of hormonal contraceptive options. Depending on the participants medical history and contraceptive preferences, they may be offered more in-depth educational videos about specific types of hormonal contraception for which they are eligible (e.g. pill, transdermal patch, intravaginal ring, injection, and implant).

Once they have completed watching the videos, participants in the intervention group will have the option of initiating one of the offered forms of birth control during the ED visit. They will only be offered medications considered low risk and for which they do not have any medical contraindications. Urine pregnancy testing will be done before any method is given. They will be able to start any contraceptive method from among those offered after their screening. Participants in the control group will be offered outpatient referral to initiate contraception, the current standard of care in our ED. All patients in both arms of the study will be given referral/follow up options for further contraceptive care.

All participants in this study will then be followed up at 1, 3, 6, and 12 months to determine continuation of contraception practices, follow up practices, satisfaction, and pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, 15-21 years old that present to the SLCH pediatric ED
* Report history of vaginal sex on the ED routine screening questionnaire
* Not currently using hormonal contraception

Exclusion Criteria:

* Pregnant
* Currently using hormonal contraception
* Foster care
* Non-English speaking
* Chief complaint of psychiatric concern, physical abuse or sexual abuse
* Triage acuity level 1 or 2 as they are likely to be too ill to participate
* Those with history of stroke, venous thromboembolism, actively being treated for cancer, or who have an organ transplant
* Too ill to participate as determined by the pediatric ED health care provider (attending physician or advanced practice nurse)
* Already participated in the study

Ages: 15 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Must be a biological female that identifies as a female.
Enrollment: 55 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Initiation of contraception in the ED using the electronic application | 12 months
  The proportion of enrolled patients that initiate contraception when offered same-day (intervention arm) compared to those that initiate contraception at follow up (the control arm) at 3 months.

SECONDARY OUTCOMES:
Delivery process related outcomes #1 | At initial encounter.
  Total length of time of the intervention beginning after consent and ending with provision of contraception, contraceptive script, or declining initiation of contraception.
Delivery process related outcomes #2 | At initial encounter.
  Subject length of stay defined by arrival time to disposition (admit or discharge) from ED.
Delivery process related outcomes #3 | At initial encounter and at follow up at 3, 6, and 12 months.
  Patient experience and satisfaction survey both directly after program and at follow up at 3, 6, and 12 months. Likert 5 point scale will be used with the following rating options strongly agree, agree, no opinion, disagree, or strongly disagree. Data will be stored in original language and in a numerical scale, with a range of 1 to 5 with 5 for the question being better experience/satisfaction. Following completion of enrollment, all data will be aggregated and analyzed to determine mean and standard deviation of all questions.
Delivery process related outcomes #4 | At initial encounter.
  Providers (doctors and nurses) experience and satisfaction survey for initial visit in ED. Likert 5 point scale will be used with the following rating options strongly agree, agree, no opinion, disagree, or strongly disagree. Data will be stored in original language and in a numerical scale, with a range of 1 to 5 with 5 for the question being better experience/satisfaction. Following completion of enrollment, all data will be aggregated and analyzed to determine mean and standard deviation of all questions.
Contraceptive continuation | At 3,6, and 12 months.
  Percentage of participants that are using hormonal contraception in the intervention group as compared to the control group at 1, 3, 6 and 12 months.
Pregnancy rates | 12 months.
  The number of participants that become pregnant within 12 months in the intervention group verses the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington Univeristy at St Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention. Reproductive Health: Teen Pregnancy. http://www.cdc.gov/teepregnancy/about/index.htm. Accessed Sept 2016.
- [Background] American College of Obstetricians and Gynecologists. Guidelines for adolescent health care. 2011; http://www.acog.org/About-ACOG/ACOG-Departments/Adolescent-Health-Care. Accessed Dec 2016.
- [Background] American Congress of Obstetricians and Gynecologists. Statement on Teen Pregnancy and Contraception. 2015; http://www.acog.org/About-ACOG/News-Room/Statements/2015/ACOG-Statement-on-Teen-Pregnancy-and-Contraception. Accessed Dec 2016.
- [Background] Committee on Adolescence. Contraception for adolescents. Pediatrics. 2014 Oct;134(4):e1244-56. doi: 10.1542/peds.2014-2299. PMID 25266430
- [Background] Healthy People 2020. Family Planning, Adolescent Health. 2014; https://www.healthypeople.gov/2020, 2017.
- [Background] Society for Adolescent Health and Medicine; Burke PJ, Coles MS, Di Meglio G, Gibson EJ, Handschin SM, Lau M, Marcell AV, Tebb KP, Urbach K. Sexual and reproductive health care: a position paper of the Society for Adolescent Health and Medicine. J Adolesc Health. 2014 Apr;54(4):491-6. doi: 10.1016/j.jadohealth.2014.01.010. No abstract available. PMID 24656535
- [Background] Chernick LS, Schnall R, Higgins T, Stockwell MS, Castano PM, Santelli J, Dayan PS. Barriers to and enablers of contraceptive use among adolescent females and their interest in an emergency department based intervention. Contraception. 2015 Mar;91(3):217-25. doi: 10.1016/j.contraception.2014.12.003. Epub 2014 Dec 12. PMID 25499588
- [Background] Chernick LS, Westhoff C, Ray M, Garcia M, Garth J, Santelli J, Dayan PS. Enhancing referral of sexually active adolescent females from the emergency department to family planning. J Womens Health (Larchmt). 2015 Apr;24(4):324-8. doi: 10.1089/jwh.2014.4994. PMID 25860108
- [Background] Ahmad FA, Jeffe DB, Plax K, Collins KK, Schechtman KB, Doerhoff DE, Garbutt J, Jaffe DM. Computerized self-interviews improve Chlamydia and gonorrhea testing among youth in the emergency department. Ann Emerg Med. 2014 Oct;64(4):376-84. doi: 10.1016/j.annemergmed.2014.01.031. Epub 2014 Mar 6. PMID 24612901
- [Background] Ahmad FA, Jeffe DB, Plax K, Schechtman KB, Doerhoff DE, Garbutt JM, Jaffe DM. Characteristics of youth agreeing to electronic sexually transmitted infection risk assessment in the emergency department. Emerg Med J. 2018 Jan;35(1):46-51. doi: 10.1136/emermed-2016-206199. Epub 2017 Aug 11. PMID 28801483